CLINICAL TRIAL: NCT03535363
Title: Phase 1 Trial of Osimertinib With Stereotactic Radiosurgery (SRS) in Patients With Brain Metastases From EGFR Positive Non-Small-Cell Lung Cancer (NSCLC)
Brief Title: Osimertinib With Stereotactic Radiosurgery (SRS) in Brain Metastases From EGFR Positive NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE3517
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: NSCLC; Non-small Cell Lung Cancer
Keywords: Osimertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Maximum Tolerated Dose of Osimertinib with standard of care (Experimental): For patients with 1-10 brain metastases, begin daily Osimeritinib 0-7 days prior to stereotactic radiosurgery (SRS), provide daily Osimeritinib concurrently with radiotherapy, followed by maintenance Osimeritinib until disease progression, withdrawal, or unacceptable toxicity. Dose Level 1: 80mg daily. Dose Level -1: 40mg daily
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Drug: Osimertinib 80mg or 40mg
  Other Names: Tagrisso

SUMMARY:
Investigating potential of controlling brain metastases in patients with EGFR positive NSCLC.

DETAILED DESCRIPTION:
In patients with EGFR positive NSCLC with 1-10 brain metastases, we are investigating whether we can control the macro brain metastases with Stereotactic Radiosurgery (SRS) and control the micro metastases with targeted agent Osimertinib and avoid whole brain radiation that could potentially lead to significant cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pathology of EGFR mutation positive NSCLC with new brain metastases.
* Ability to care for self and ability to walk 50% of waking hours (ECOG Performance Status of 0-2)
* 1-10 brain metastases with intra-cranial brain metastasis must measure 3cm or less in the greatest dimension.
* Hemoglobin ≥9 g/dL, White Blood Count Absolute ≥3.0 x 10^9/L, Granulocyte count ≥1.5 x 10^9/L, and platelet count ≥100 x 10^9/L
* Serum Bilirubin ≤ 1.5 x upper limit of normal (ULN)
* AST and/or ALT ≤ 2 ULN (≤ 5 x ULN when clearly attributable to liver metastases)
* Serum creatinine ≤ 1.5 ULN or calculated creatinine clearance > 60ml/min
* For women of childbearing potential-Negative pregnancy test within one week prior to start of therapy.
* For all sexually active male and female patients of reproductive potential, employ two methods of highly effective and acceptable forms of contraception throughout the study and for 120 days following the final dose of osimertinib.

Exclusion Criteria:

* Patients with leptomeningeal metastases documented by MRI or cerebrospinal fluid (CSF).
* Significant intratumoral or peritumoral hemorrhage
* Brain metastases within 5 mm of the optic chiasm or optic nerve
* Brainstem metastases
* Gastrointestinal disorders with diarrhea as a major symptom
* Clinically significant or uncontrolled cardiac disease (NYHA functional classification of 3 or 4)
* Pre-existing interstitial lung disease or pneumonitis
* Unable to undergo brain MRI
* HIV or Hepatitis B or C
* Prior treatments must be resolved to an asymptomatic state at time of enrollment
* Medical conditions that could cause safety risks
* Currently receiving investigational cancer therapy.
* Mean QT interval corrected heart rate (QTc)≥470ms calculated from 3 EKGs
* Left Ventricular Ejection Fraction (LVEF) ≤ 50%
* Use of strong CYP3A inhibitors
* Use of strong CYP3A4 inducers
* Use of potent CYP2C8 inhibitors
* Hypersensitivity to osimertinib or any of its ingredients
* corneal ulceration
* pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Osimertinib with (SRS) | 4 weeks
  To determine the safety, tolerability and maximum tolerated dose of Osimertinib, when administered in combination with SRS in patients with EGFR positive NSCLC with brain metastases.

SECONDARY OUTCOMES:
Number of patients with progression free survival | 6 months
  To assess the six-month intra-cranial and extra-cranial progression-free survival (PFS-6) in patients with EGFR positive NSCLC brain metastases treated with Osimertinib and SRS (PFS is defined as the time from clinical registration to intra-or extra-cranial tumor progression or death)
Length of overall survival | 2 years
  To assess the overall survival (OS) in patients with EGFR positive NSCLC Brain Metastases treated with Osimertinib and SRS
Difference in outcome vs. standard of care | 2 years
  To compare results of our clinical trial to patients with EGFR positive NSCLC with brain metastases treated with SRS alone (1-10 brain Metastases)
Intra-cranial and Extra-cranial Overall Response Rate (ORR) | 6 months
  To assess Overall response rate (ORR) both intracranial and extracranial, defined as the proportion of patients with a best overall confirmed response of complete response (CR) or partial response (PR) in the whole body as assessed per RECIST 1.1 by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Glen Stevens, DO, PhD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Maimi Cancer Institute - Baptist Health South Florida, Miami, Florida
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio